CLINICAL TRIAL: NCT04183140
Title: Comparation of Transulnar Versus Transradial Approach for Primary Percutaneous Coronary Intervention in Patients With ST-elevated Myocardial Infarction in Terms of Procedure Complications and In-hospital Cardiac Outcomes
Brief Title: Comparison of Radial and Ulnar Artery Intervention in Patients With ST Elevated Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Kahraman Cosansu, Principal Investigator, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SEAH
Record Dates: First submitted 2019-11-15; First posted 2019-12-03 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: ST Elevated Myocardial Infarction
Keywords: Complication; Primary Percutaneus Coronary Intervention; Radial Artery; Ulnar Artery
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Patients admitted with STEMI at the cardiology department and admitted to the catheter laboratory for primary percutaneous coronary intervention will be included in the study. There will be two groups in the study.In the first group, patients treated with transulnar access will be included. In the second group, patients using transradial access will be included. Patients will be treated by the same operator respectively. Peri-procedural data and in-hospital cardiac outcome data of patients in both groups will be recorded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transradial (Active Comparator): Transradial intervention
  Interventions: Procedure: primary percutaneous coronary intervention
- Transulnar (Active Comparator): Transulnar intervention
  Interventions: Procedure: primary percutaneous coronary intervention

INTERVENTIONS:
Procedure: primary percutaneous coronary intervention — primary percutaneous coronary intervention via transulnar or transradial access

SUMMARY:
In the literature, there are no studies comparing these two pathways in ST elevation myocardial infarction (STEMI). In this patient group, it will be investigated whether transulnar intervention causes similar or less complications than transradial intervention, and whether it provides superiority or similarity in terms of outcomes.

DETAILED DESCRIPTION:
The transulnar approach is known as an alternative procedure for transradial coronary angiography due to its safety and applicability. For cardiologists, experienced in trans-ulnar access, this access zone is comfortable to use. Because less spasm is developing. In addition, no significant difference was found between the transradial and transulnar routes in terms of other complications.In the literature, there are no studies comparing these two pathways in ST elevation myocardial infarction (STEMI). In this patient group, it will be investigated whether transulnar intervention causes similar or less complications than transradial intervention, and whether it provides superiority or similarity in terms of outcomes.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age
* admitted for primary percutaneous intervention
* either of these two routes has not been used in the last week
* a sufficient pulse at both routes

Exclusion Criteria:

* cardiogenic shock
* stent thrombosis
* the use of either of these two arteries in the last 1 week
* either of these arteries can not be pulsed or very weak pulsed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Complication rate | 1 day
  Major and minor neurovascular events (access related) of the arm including pain/motor paralysis/paresthesia, hematoma, pseudoaneurysm, artery spasm, arterial occlusion
in-hospital cardiac outcomes | 1 week
  the incidence of death, myocardial infarction (MI), urgent target lesion revascularization (TLR), acute heart failure as major adverse cardiac events (MACEs) within the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Kahraman Cosansu, Principal Investigator — Sakarya University
Locations (1):
- Sakarya University Education and Research Hospital, Sakarya, TR, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roghani-Dehkordi F, Mansouri R, Khosravi A, Mahaki B, Akbarzadeh M, Kermani-Alghoraishi M. Transulnar versus transradial approach for coronary angiography and angioplasty: Considering their complications. ARYA Atheroscler. 2018 May;14(3):128-131. doi: 10.22122/arya.v14i3.1586. PMID 30349575
- [Background] Bi X, Wang Q, Liu D, Gan Q, Liu L. Is the Complication Rate of Ulnar and Radial Approaches for Coronary Artery Intervention the Same? Angiology. 2017 Nov;68(10):919-925. doi: 10.1177/0003319717703226. Epub 2017 Apr 7. PMID 28387125
- [Background] Dahal K, Rijal J, Lee J, Korr KS, Azrin M. Transulnar versus transradial access for coronary angiography or percutaneous coronary intervention: A meta-analysis of randomized controlled trials. Catheter Cardiovasc Interv. 2016 Apr;87(5):857-65. doi: 10.1002/ccd.26221. Epub 2015 Sep 2. PMID 26332022
- [Background] Geng W, Fu X, Gu X, Jiang Y, Fan W, Wang Y, Li W, Xing K, Liu C. Safety and feasibility of transulnar versus transradial artery approach for coronary catheterization in non-selective patients. Chin Med J (Engl). 2014;127(7):1222-8. PMID 24709170